CLINICAL TRIAL: NCT04347551
Title: Motor Performance of Asymptomatic and Chronic Neck Pain Participants Pre- and Post-spinal Manipulation Using an Eye and Head Movement Fitts' Task
Brief Title: The Effects of Spinal Manipulation on Performance on Neck Pain Patients During a Fitts' Task
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Geoff Gelley, PhD Candidate, University of Manitoba
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B2020:010
Record Dates: First submitted 2020-04-08; First posted 2020-04-15 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Chronic Neck Pain
Keywords: Manipulation, Spinal; Fitts' Task; Motor Performance
MeSH Terms: interventions — Manipulation, Spinal

STUDY DESIGN:
Intervention Model Description: This is an observational within-subjects design that involves a pre/post cervical spine manipulation intervention on participants (n=20) with chronic neck pain and asymptomatic controls (n=20). All participants will complete an eye movement and head movement Fitts' task before and after cervical spine manipulation to identify any changes in eye and head movement time, eye and head peak velocity, and time to peak eye and head velocity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye movement Fitts' task (Experimental): High velocity/low amplitude cervical spine manipulation applied to chronic neck pain and asymptomatic participants.
  Interventions: Other: High velocity/low amplitude cervical spine manipulation
- Head movement Fitts' task (Active Comparator): High velocity/low amplitude cervical spine manipulation applied to chronic neck pain and asymptomatic participants.
  Interventions: Other: High velocity/low amplitude cervical spine manipulation

INTERVENTIONS:
Other: High velocity/low amplitude cervical spine manipulation — The participants will receive a single cervical spine rotary manipulation to the previously identified palpable cervical segmental fixation. During the performance of the manipulation, the supine participant will rest their arms at the sides of their body. Next, the index finger of the chiropractor's contact hand will be placed on the lamina of the restricted cervical segment. The chiropractor will then rotate the participant's head contralaterally until the barrier of the cervical segments volitional end range is reached. The chiropractor's other hand will be placed behind the participant's head to induce gentle neck rotation contralateral to the chiropractor's thrusting hand. The chiropractor will deliver a manual thrust, with the thrust vector directed towards the participant's opposite eye.
  Other Names: Cervical manipulation; Neck manipulation; Cervical adjustment; Neck adjustment

SUMMARY:
The objective of this study is to quantify motor performance, this study will use an eye movement Fitts' task to examine the effects of cervical spine manipulation on participants with chronic neck pain and the subsequent changes to saccade movement time. This study will also include a head movement Fitts' task which has previously reported a reduction in head movement time in chronic neck pain participants after cervical spine manipulation.

This is an observational within-subjects design that involves a pre/post cervical spine manipulation intervention on participants (n=20) with chronic neck pain and asymptomatic controls (n=20). All participants will complete an eye movement and head movement Fitts' task before and after cervical spine manipulation to identify any changes in saccade and head movement time, saccade and head peak velocity, and time to peak saccade and head velocity.

DETAILED DESCRIPTION:
The purpose of this study is to measure the effects of cervical spine manipulation on the motor performance of participants with and without chronic neck pain.

The objective of this pre/post design study is to apply spinal manipulation of the cervical spine to participants with chronic neck pain and participants who are asymptomatic for neck pain, and to measure the subsequent changes of movement time of the eyes during an eye movement Fitts' task using eye-tracker technology.

This study will also include a head movement Fitts' task, which has been previously shown to identify a reduction in head movement time in participants after receiving cervical spine manipulation. The head movement task, which has a biomechanical basis, will serve as a comparator to the eye movement task, which has a neurophysiologic basis. Changes in head and eye movement time are both measures of motor performance.

The hypothesis for the eye movement Fitts' task, is that the eye movement time will be increase with larger distances between targets and will not be affected by changes in target width. It is anticipated that the eye movement time will reduce in the neck pain group following spinal manipulation in comparison to the asymptomatic group. We hypothesize that during the head movement task, symptomatic participants will experience a decrease in head movement time as compared to the asymptomatic group after spinal manipulation. We further hypothesize that head movement time will be increase with larger target distances and smaller target widths.

ELIGIBILITY:
Participants with neck pain:

Inclusion criteria

* Between the ages of 18 and 40
* Neck pain for at least 3 months
* Palpable spinal segmental fixations at C1-7
* Neck pain must be reproducible by neck movements and/or provocative
* Normal or corrected-to-normal vision

Exclusion criteria

* Contraindications to spinal manipulation
* Can't be calibrated during the eye movement Fitts task (excluded from eye movement test only)
* Progressive neurologic deficits
* Cervical spine trauma or surgery
* Infection, tumor, osteoporosis, inflammatory spondyloarthropathy, spinal fracture, and a history of vestibular/inner ear dysfunction
* Diagnosed with an autonomic disorder such as Horner's syndrome
* Any current ocular and/or retinal disease, Diabetes, a history of head trauma
* Currently using opioids, recreational drugs or have a history of substance abuse

Asymptomatic participants:

Inclusion criteria

* Between the ages of 18 and 40
* No neck pain for at least 3 months
* Palpable spinal segmental fixations at C1-7
* Normal or corrected-to-normal vision

Exclusion criteria

* Contraindications to spinal manipulation
* Can't be calibrated during the eye movement Fitts task (excluded from eye movement test only)
* Progressive neurologic deficits
* Cervical spine trauma or surgery
* Infection, tumor, osteoporosis, inflammatory spondyloarthropathy, spinal fracture, and a history of vestibular/inner ear dysfunction
* Diagnosed with an autonomic disorder such as Horner's syndrome
* Any current ocular and/or retinal disease, Diabetes, a history of head trauma
* Currently using opioids, recreational drugs or have a history of substance abuse

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Change in eye (saccade) movement time | Change from baseline saccade movement time immediately following cervical spine manipulation.
  Eye (saccade) movement time (milliseconds), which is the time between saccade onset and offset while moving from central circle to the target.
Change in head movement time | Change from baseline head movement time immediately following cervical spine manipulation.
  Head movement time (milliseconds) is the time required to move the cursor from the central circle to the target.

SECONDARY OUTCOMES:
Change in saccade peak velocity | Change from baseline saccade peak velocity immediately following cervical spine manipulation.
  Peak of the velocity amplitude (meters/second) in the horizontal movement direction
Change in time to peak saccade velocity | Change from baseline time to peak velocity immediately following cervical spine manipulation.
  Measured as the time (milliseconds) from the onset of velocity to its peak amplitude
Change in head peak velocity | Change from baseline head peak velocity immediately following cervical spine manipulation.
  Measured as the peak of the velocity amplitude (meters/second) of the cursor moving in the horizontal plane
Change in time to peak head velocity | Change from baseline time to peak head velocity immediately following cervical spine manipulation.
  The time (milliseconds) to peak velocity will be measured as the time from the onset of velocity to its peak amplitude.

OTHER OUTCOMES:
Change in Visual analog scale (VAS) score | Change from baseline Visual Analog Scale (VAS) score immediately following cervical spine manipulation.
  100 mm visual analog scale (VAS) to score their pain intensity
The Neck Disability Index (NDI) score | Baseline prior to cervical spine manipulation
  To quantify neck disability related to work and physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Gelley, DC, MSc, Principal Investigator — University of Manitoba
Locations (1):
- Gelley Chiropractic Office, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
I will be sharing processed and analyzed data.
  The results of this study will be prepared for dissemination first at relevant clinical and scientific conferences. Subsequently, this work will be submitted to a peer reviewed journal for consideration of publication. Datasets will be deposited in the University of Manitoba's Dataverse.
  The data collected during this study may be shared in an anonymized or de-identified form with academic journals for publication purposes or other researchers according to international guidelines. The data may also be stored by the academic journal under an open access policy in which case it may be used by other researchers for further data analysis and research purposes. Before publishing/sharing any data, it will be reviewed with the Research Ethics Board or oversight committee to ensure full compliance with privacy legislation.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Uncertain as research has been placed on hold due to the COVID-19 pandemic.
Access Criteria: Datasets will be deposited in the University of Manitoba's Dataverse. Dataverse is an open source web application to share, preserve, cite, explore, and analyze research data.
URL: https://dataverse.org

REFERENCES:
- [Background] Bialosky JE, George SZ, Horn ME, Price DD, Staud R, Robinson ME. Spinal manipulative therapy-specific changes in pain sensitivity in individuals with low back pain (NCT01168999). J Pain. 2014 Feb;15(2):136-48. doi: 10.1016/j.jpain.2013.10.005. Epub 2013 Oct 27. PMID 24361109
- [Background] Boal RW, Gillette RG. Central neuronal plasticity, low back pain and spinal manipulative therapy. J Manipulative Physiol Ther. 2004 Jun;27(5):314-26. doi: 10.1016/j.jmpt.2004.04.005. PMID 15195039
- [Background] Fitts PM. The information capacity of the human motor system in controlling the amplitude of movement. 1954. J Exp Psychol Gen. 1992 Sep;121(3):262-9. doi: 10.1037//0096-3445.121.3.262. No abstract available. PMID 1402698
- [Background] Fitts PM, Radford BK. Information capacity of discrete motor responses under different cognitive sets. J Exp Psychol. 1966 Apr;71(4):475-82. doi: 10.1037/h0022970. No abstract available. PMID 5909070
- [Background] Flor H, Braun C, Elbert T, Birbaumer N. Extensive reorganization of primary somatosensory cortex in chronic back pain patients. Neurosci Lett. 1997 Mar 7;224(1):5-8. doi: 10.1016/s0304-3940(97)13441-3. PMID 9132689
- [Background] Fryer G, Morris T, Gibbons P. Paraspinal muscles and intervertebral dysfunction: part one. J Manipulative Physiol Ther. 2004 May;27(4):267-74. doi: 10.1016/j.jmpt.2004.02.006. PMID 15148466
- [Background] Gay CW, Robinson ME, George SZ, Perlstein WM, Bishop MD. Immediate changes after manual therapy in resting-state functional connectivity as measured by functional magnetic resonance imaging in participants with induced low back pain. J Manipulative Physiol Ther. 2014 Nov-Dec;37(9):614-27. doi: 10.1016/j.jmpt.2014.09.001. Epub 2014 Oct 3. PMID 25284739
- [Background] Gelley GM, Passmore SR, MacNeil BJ. Acceleration of clinician hand movements during spinal manipulative therapy. Man Ther. 2015 Apr;20(2):342-8. doi: 10.1016/j.math.2014.10.010. Epub 2014 Oct 31. PMID 25458144
- [Background] George SZ, Bishop MD, Bialosky JE, Zeppieri G Jr, Robinson ME. Immediate effects of spinal manipulation on thermal pain sensitivity: an experimental study. BMC Musculoskelet Disord. 2006 Aug 15;7:68. doi: 10.1186/1471-2474-7-68. PMID 16911795
- [Background] Gross A, Miller J, D'Sylva J, Burnie SJ, Goldsmith CH, Graham N, Haines T, Bronfort G, Hoving JL; COG. Manipulation or mobilisation for neck pain: a Cochrane Review. Man Ther. 2010 Aug;15(4):315-33. doi: 10.1016/j.math.2010.04.002. Epub 2010 May 26. PMID 20510644
- [Background] Gyer G, Michael J, Inklebarger J, Tedla JS. Spinal manipulation therapy: Is it all about the brain? A current review of the neurophysiological effects of manipulation. J Integr Med. 2019 Sep;17(5):328-337. doi: 10.1016/j.joim.2019.05.004. Epub 2019 May 9. PMID 31105036
- [Background] Haavik-Taylor H, Murphy B. Cervical spine manipulation alters sensorimotor integration: a somatosensory evoked potential study. Clin Neurophysiol. 2007 Feb;118(2):391-402. doi: 10.1016/j.clinph.2006.09.014. Epub 2006 Nov 29. PMID 17137836
- [Background] Haavik H, Murphy B. Subclinical neck pain and the effects of cervical manipulation on elbow joint position sense. J Manipulative Physiol Ther. 2011 Feb;34(2):88-97. doi: 10.1016/j.jmpt.2010.12.009. PMID 21334540
- [Background] Haavik H, Murphy B. The role of spinal manipulation in addressing disordered sensorimotor integration and altered motor control. J Electromyogr Kinesiol. 2012 Oct;22(5):768-76. doi: 10.1016/j.jelekin.2012.02.012. Epub 2012 Apr 6. PMID 22483612
- [Background] Haavik Taylor H, Murphy B. The effects of spinal manipulation on central integration of dual somatosensory input observed after motor training: a crossover study. J Manipulative Physiol Ther. 2010 May;33(4):261-72. doi: 10.1016/j.jmpt.2010.03.004. PMID 20534312
- [Background] Haneline MT, Cooperstein R, Young M, Birkeland K. Spinal motion palpation: a comparison of studies that assessed intersegmental end feel vs excursion. J Manipulative Physiol Ther. 2008 Oct;31(8):616-26. doi: 10.1016/j.jmpt.2008.09.007. PMID 18984245
- [Background] Herzog W. The biomechanics of spinal manipulation. J Bodyw Mov Ther. 2010 Jul;14(3):280-6. doi: 10.1016/j.jbmt.2010.03.004. PMID 20538226
- [Background] Lersa LB, Stinear CM, Lersa RA. The relationship between spinal dysfunction and reaction time measures. J Manipulative Physiol Ther. 2005 Sep;28(7):502-7. doi: 10.1016/j.jmpt.2005.07.007. PMID 16182024
- [Background] Marchand AA, Cantin V, Murphy B, Stern P, Descarreaux M. Is performance in goal oriented head movements altered in patients with tension type headache? BMC Musculoskelet Disord. 2014 May 26;15:179. doi: 10.1186/1471-2474-15-179. PMID 24884672
- [Background] Passmore SR, Burke JR, Good C, Lyons JL, Dunn AS. Spinal manipulation impacts cervical spine movement and fitts' task performance: a single-blind randomized before-after trial. J Manipulative Physiol Ther. 2010 Mar-Apr;33(3):189-92. doi: 10.1016/j.jmpt.2010.01.007. PMID 20350671
- [Background] Passmore SR, Descarreaux M. Performance based objective outcome measures and spinal manipulation. J Electromyogr Kinesiol. 2012 Oct;22(5):697-707. doi: 10.1016/j.jelekin.2012.02.005. Epub 2012 Mar 8. PMID 22406070
- [Background] Pickar JG, Bolton PS. Spinal manipulative therapy and somatosensory activation. J Electromyogr Kinesiol. 2012 Oct;22(5):785-94. doi: 10.1016/j.jelekin.2012.01.015. Epub 2012 Feb 19. PMID 22349622
- [Background] Pickar JG, Wheeler JD. Response of muscle proprioceptors to spinal manipulative-like loads in the anesthetized cat. J Manipulative Physiol Ther. 2001 Jan;24(1):2-11. doi: 10.1067/mmt.2001.112017. PMID 11174689
- [Background] Reed WR, Cranston JT, Onifer SM, Little JW, Sozio RS. Decreased spontaneous activity and altered evoked nociceptive response of rat thalamic submedius neurons to lumbar vertebra thrust. Exp Brain Res. 2017 Sep;235(9):2883-2892. doi: 10.1007/s00221-017-5013-5. Epub 2017 Jul 7. PMID 28687855
- [Background] Reed WR, Liebschner MA, Sozio RS, Pickar JG, Gudavalli MR. Neural Response During a Mechanically Assisted Spinal Manipulation in an Animal Model: A Pilot Study. J Nov Physiother Phys Rehabil. 2015 Sep;2(2):20-27. doi: 10.17352/2455-5487.000021. Epub 2015 Apr 6. PMID 26618202
- [Background] Reed WR, Long CR, Kawchuk GN, Pickar JG. Neural responses to the mechanical parameters of a high-velocity, low-amplitude spinal manipulation: effect of preload parameters. J Manipulative Physiol Ther. 2014 Feb;37(2):68-78. doi: 10.1016/j.jmpt.2013.12.004. Epub 2014 Jan 3. PMID 24387888
- [Background] Sillevis R, Cleland J, Hellman M, Beekhuizen K. Immediate effects of a thoracic spine thrust manipulation on the autonomic nervous system: a randomized clinical trial. J Man Manip Ther. 2010 Dec;18(4):181-90. doi: 10.1179/106698110X12804993427126. PMID 22131791
- [Background] Smith DL, Dainoff MJ, Smith JP. The effect of chiropractic adjustments on movement time: a pilot study using Fitts Law. J Manipulative Physiol Ther. 2006 May;29(4):257-66. doi: 10.1016/j.jmpt.2006.03.009. PMID 16690379
- [Background] Stochkendahl MJ, Christensen HW, Hartvigsen J, Vach W, Haas M, Hestbaek L, Adams A, Bronfort G. Manual examination of the spine: a systematic critical literature review of reproducibility. J Manipulative Physiol Ther. 2006 Jul-Aug;29(6):475-85, 485.e1-10. doi: 10.1016/j.jmpt.2006.06.011. PMID 16904495
- [Background] Treleaven J. Sensorimotor disturbances in neck disorders affecting postural stability, head and eye movement control. Man Ther. 2008 Feb;13(1):2-11. doi: 10.1016/j.math.2007.06.003. Epub 2007 Aug 16. PMID 17702636